CLINICAL TRIAL: NCT02855073
Title: A Randomized, Single-blind, Phase II Clinical Trial to Compare ReJoinTM (Autologous Adipose-derived Mesenchymal Progenitor Cells)to Sodium Hyaluronate Injection for the Patients With Knee Osteoarthritis Cartilage Defects
Brief Title: Clinical Trial to Compare ReJoinTM to Sodium Hyaluronate Injection for Knee Osteoarthritis Cartilage Defects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CBMG-ReJoinTM-CL-1.0
Record Dates: First submitted 2016-07-08; First posted 2016-08-04 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Defect of Articular Cartilage; Knee Osteoarthritis
Keywords: adipose-derived mesenchymal progenitor cells; Artz
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReJoinTM Group (Experimental): Subjects in this Group will receive ReJoinTM injections on day 1 and day 22, and Sodium Hyaluronate injection on day 8 and day 15.
  Interventions: Biological: ReJoinTM
- Sodium Hyaluronate Group (Active Comparator): subjects in this group will receive Sodium Hyaluronate injections on day 1, 8, 15, 22.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Biological: ReJoinTM — adipose derived mesenchymal progeinitor cells
  Other Names: adipose derived mesenchymal progenitor cells
  Arms: ReJoinTM Group
Drug: Sodium Hyaluronate — Sodium Hyaluronate Injection
  Other Names: Artz
  Arms: Sodium Hyaluronate Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ReJoinTM for the Knee Osteoarthritis patients with Cartilage Defects comparing to Sodium Hyaluronate Injection.

DETAILED DESCRIPTION:
This is a randomized, single-blind,phase II clinical trial.

At least 28 subjects who are with a clinical diagnosis of knee osteoarthritis cartilage defects will be randomly distributed 1:1 to the treatment group or the control group after signing the ICF and screening tests.The treatment will accept ReJoinTM at the first and fourth week,and Sodium Hyaluronate Injection at the second and third week.The control group will accept Sodium Hyaluronate Injection weekly ,and four injections in total.The duration of the therapy is 48 weeks.

In addition, external control will be added if necessary.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, KOA couse ≤ 10 years
* Kellgren-Lawrence Ⅰ-Ⅲ
* VAS core >6， more than 4 months
* Signed informed consent from the subject
* cartilage defect 2-6cm2

Exclusion Criteria:

* Pregnancy test positive.
* Subject infected with hepatitis C, HIV or syphilis.
* Subject enrolled in any other cell therapy studies within the past 30 days.
* Subject deemed to be not suitable for the study by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC scores | 48 weeks
  WOMAC scoring will be performed 48 weeks after the first injection

SECONDARY OUTCOMES:
VAS scores | 0 day、8 weeks、24 weeks、36 weeks and 48 weeks
  VAS scoring will be performed 8 weeks、24 weeks、36 weeks and 48 weeks after the first injection
SF-36 scores | 0 day、8 weeks、24 weeks、 36 weeks and 48 weeks
  SF-36 scoring will be performed 8 weeks、24 weeks、36 weeks and 48 weeks after the first injection
Outbridge scoring | 1 day and 24 weeks
  Outbridge scoring will be performed 24 weeks after the first injection under arthroscopy
CRP | 0 day、8 weeks、24 weeks、 36 weeks and 48 weeks
  Serum CRP levels will be tested 8 weeks、24 weeks、36 weeks and 48 weeks after the first injection
Cartilage defect size | 0 day and 24 weeks
  Cartilage defect size will be measured at 24 weeks after the first injection
Cartilage volume | 0 day and 24 weeks
  Cartilage volume will be measured at 24 weeks after first injection

CONTACTS AND LOCATIONS:
Overall Officials: You Wang, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qiao Z, Tang J, Yue B, Wang J, Zhang J, Xuan L, Dai C, Li S, Li M, Xu C, Dai K, Wang Y. Human adipose-derived mesenchymal progenitor cells plus microfracture and hyaluronic acid for cartilage repair: a Phase IIa trial. Regen Med. 2020 Jan;15(1):1193-1214. doi: 10.2217/rme-2019-0068. Epub 2020 Feb 11. PMID 32043426